CLINICAL TRIAL: NCT03955172
Title: Efficiency of Everolimus for the Treatment of Kidney Transplanted Patients Presenting a Missing Self-induced Natural Killer Cells Mediated (NK-mediated) Rejection
Brief Title: Efficiency of Everolimus for the Treatment of Kidney Transplanted Patients Presenting a Missing Self-induced NK-mediated Rejection
Acronym: STARR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0706
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: Missing self; NK cells; Rejection; mTOR inhibitors; Kidney transplanted patients
MeSH Terms: conditions — Rejection, Psychology | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Everolimus (Experimental)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Patients will received everolimus (CERTICAN), oral form, at the necessary dose to obtain trough levels between 6 and 8 ng/ml, during 6 months. Everolimus will replace the anti-proliferative drug they have before (azathioprine or mycophenolic acid). Everolimus will be associated with corticosteroids (prednisolone) and a calcineurin inhibitor (tacrolimus or cyclosporin).

SUMMARY:
Background:

Long-term success of organ transplantation is limited by the inexorable loss of graft function due to rejection. Prevalent dogma defends that allograft rejection is exclusively mediated by the adaptive immune system: T cells are responsible for cellular rejections and B cells producing Donor Specific Antibodies (DSA) are responsible for humoral rejection. Recently, we demonstrated that innate NK cells could be implicated in the generation of chronic vascular rejections lesions by sensing the absence of expression of self Major Histocompatibility Complex (MHC) class I molecules ("missing self") on graft endothelial cells with their Killer cell immunoglobulin-like (KIR) receptors. Using human in vitro and murine in vivo models, we also showed that Mammalian Target Of Rapamycin (mTOR) inhibitors could efficiently prevent this new kind of rejection.

Objective:

The aim of our project is therefore to test in a cohort of kidney transplanted patients the efficiency of mTOR inhibitors to treat this new kind of rejection

Methods:

A cohort of 20 kidney transplant patients with a missing self on their graft responsible for a NK-mediated rejection will be established prospectively. An mTOR inhibitor will be introduced in these patients for 6 months in association with a calcineurin inhibitor and corticosteroids. Graft function, histological lesions and NK activability will be monitored following this modification of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged > 18 years
* Kidney transplanted patient
* Having microvascular inflammation lesion on his graft biopsy associated to mild chronic lesions
* In absence of donor specific antibodies
* In presence of a missing self

Exclusion Criteria:

* Proteinuria/urinary creatinin > 100 mg/mmol
* Antecedent of poor tolerance or hypersensibility to everolimus or sirolimus
* Severe chronic lesions
* Presence of donor specific antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2027-12-03 (Estimated); Study Completion 2027-12-03 (Estimated)

PRIMARY OUTCOMES:
Change in Estimated glomerular filtration rate | 6 months after start of Everolimus treatment
  Glomerular filtration rate will be estimated by Chronic Kidney Disease - Epidemiology CollaborationI (CKD-EP) equation.
  Outcome evaluation at 6 months after everolimus treatment introduction (at D0) compared to baseline (between 15 and 30 days before D0).

SECONDARY OUTCOMES:
Change in the severity of rejection lesions on allograft biopsy | 6 months after start of Everolimus treatment
  Evolution of microvascular inflammation and chronic glomerular and vascular lesions graded according to Banff 2013 classification.
  Outcome evaluation at 6 months after everolimus treatment introduction (at D0) compared to baseline (between 15 and 30 days before D0).
Change in NK cell activability | 6 months after start of Everolimus treatment
  Nk cell activability will be measured by looking at the expression of activation markers (CD107a and MIP1B) on circulating NK cells by flow cytometry.
  Outcome evaluation at 6 months after everolimus treatment introduction (at D0) compared to baseline (between 15 and 30 days before D0).
Change in proteinuria | 6 months after start of Everolimus treatment
  Calculation of proteinuria/urinary creatinin index. Outcome evaluation at 6 months after everolimus treatment introduction (at D0) compared to baseline (between 15 and 30 days before D0).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de transplantation, néphrologie et immunologie clinique, Hôpital Edouard Herriot (HCL), Lyon, France